CLINICAL TRIAL: NCT04766528
Title: Effect of Dietary Composition on the Gut Microbiota / Endocannabinoidome Axis in Response to Maximal Aerobic Exercise
Brief Title: Effect of Diet on the Microbiota / Endoccanabinoidome Axis in Response to Physical Activity
Acronym: PerOME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2019-005
Record Dates: First submitted 2021-02-19; First posted 2021-02-23 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2019-10

CONDITIONS: Diet Habit; Microbial Colonization; Activity, Motor
Keywords: Microbiome; Endocannabinoids
MeSH Terms: conditions — Feeding Behavior; Communicable Diseases; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mediterannen diet (Experimental): The MED diet was abundant in fiber, micronutrients and plant-based proteins. The diet was rich in essential FA like monounsaturated fatty acids (MUFA) and n-3.
  Interventions: Other: 3 maximal aerobic tests
- Canadian diet (Experimental): The NAM diet had a high content in saturated fatty acids (SFA) and simple sugar and was low in fiber.
  Interventions: Other: 3 maximal aerobic tests

INTERVENTIONS:
Other: 3 maximal aerobic tests — Maximal aerobic tests will be performed before diet intervention, after the first diet and after the second diet

SUMMARY:
Both the endocannabinoid system and the microbiome are highly conditioned by nutrition and physical activity, and have an interdependent, bidirectional relationship. We suggest studying the interleaving between the endocannabinoidome-microbiome axis and host metabolism under the combined effect of a diet and physical activity. More specificly, we will study the link between the impact of the diet on the intestinal microbiome and the endocannabinoid reaction after intense exercise.

DETAILED DESCRIPTION:
Aims of the study are to compare the impacts of two short 7-day contrasted nutritional interventions (the Mediterranean diet (MED) and the Canadian diet (CAN)) on blood metabolites (endocannabinoids) after a maximal aerobic test. A 3 weeks washout between the two diets is planned. Gut microbiome at each test will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* women
* 20-30 years old
* healthy
* jogging >1h/week and >3h/week of physical activity
* bmi 18.5-25

Exclusion Criteria:

* postmenopausal, pregnancy or lactation
* pathology or medication
* smoking
* more than 7 alcohol consumption/week
* food allergy, food intolerance or food aversion
* important weight change in the last 6 months
* antibiotics in the last 3 months
* night worker
* pathologies

Ages: 20 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2019-09-06 (Actual); Primary Completion 2019-11-14 (Actual); Study Completion 2019-11-14 (Actual)

PRIMARY OUTCOMES:
Endocannabinoid level post physical activity | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Institut sur la nutrition et les aliments fonctionnels, Québec, Canada

IPD SHARING:
Plan to Share IPD: No